CLINICAL TRIAL: NCT06398626
Title: A Multi-Center, Prospective, Non-Interventional Study of Real-World Effectiveness of Etrasimod in Patients With Ulcerative Colitis (ENDEAVOUR-UC)
Brief Title: An Observational Study of Etrasimod in Adult Patients With Moderate to Severe Ulcerative Colitis
Acronym: ENDEAVOUR-UC
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C5041047; ENDEAVOUR-UC (Other: Alias Study Number)
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients with ulcerative colitis taking etrasimod
  Interventions: Drug: Etrasimod

INTERVENTIONS:
Drug: Etrasimod — As provided in real world practice

SUMMARY:
The purpose of this observational study is to learn about the effects of etrasimod as a treatment for adult patients with moderate to severe ulcerative colitis. Patients will be treated according to standard of care and will only be included in the study if etrasimod is the best treatment of choice according to the physician and they have not previously taken etrasimod.

All patients will be prescribed etrasimod according to standard of care. Tests and doctor visits will be conducted according to standard of care with the exception of health questionnaires about ulcerative colitis symptoms. These questionnaires will be completed by patients at various timepoints during the study using their mobile phone, tablet, or computer.

The study is 52 weeks with 28 days of safety follow up. The effects of etrasimod will be analyzed for each patient comparing their disease activity prior to the start of etrasimod.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and < 65 years at baseline
2. Patients with confirmed diagnosis of UC who are prescribed etrasimod for moderately to severely active UC
3. Evidence of a personally signed and dated ICD indicating that the patient (or a legally acceptable representative)has been informed of all pertinent aspects of the study

Exclusion Criteria:

1. The presence of clinical findings suggestive of Crohn's disease
2. Severe extensive colitis evidenced by:

   1. Physician judgement that the patient is likely to require hospitalization for medical or surgical intervention of any kind for UC (e.g., colectomy) within 12 weeks
   2. Current evidence of acute severe UC, fulminant colitis, or toxic megacolon
3. Patients with a stoma or planned UC surgical intervention requiring hospitalization
4. Prior/Concomitant Therapy:

   1. Any previous exposure to etrasimod, including participation in the etrasimod clinical program
   2. Any co-medication with one of the following conventional therapies: methotrexate or a thiopurine (azathioprine, mercaptopurine, or tioguanine)
   3. Any co-medication with one of the following advanced therapies for UC: biologics (a TNF, integrin or cytokine antagonist; JAKi [filgotinib, tofacitinib, or upadacitinib]) or with any other S1P receptor modulator
5. Unwillingness or inability to download the web-based tool to complete ePROs on a personal device or not capable of using the web-based tool
6. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible patients can be included in this study if their physician makes a clinical decision to treat them with etrasimod, as defined by the United States etrasimod prescribing information and independent from the decision to enroll the patient in this study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-07-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with symptomatic remission | Week 12
  Symptomatic remission is defined as partial Modified Mayo Score (pMMS) stool frequency subscore (SFS) = 0 (or = 1 with a ≥ 1-point decrease from baseline) and (RBS) rectal bleeding subscore = 0

SECONDARY OUTCOMES:
Proportion of patients with symptomatic remission | Weeks 24, 36, 52
  Symptomatic remission is defined as partial Modified Mayo Score (pMMS) stool frequency subscore (SFS) = 0 (or = 1 with a ≥ 1-point decrease from baseline) and (RBS) rectal bleeding subscore = 0
Proportion of patients with symptomatic response | Weeks 12, 24, 36, 52
  Symptomatic response defined as a decrease from baseline ≥ 30% in pMMS composite RBS and SFS
Proportion of patients with symptomatic response | Weeks 12, 24, 36, 52
  Symptomatic response defined as a decrease from baseline ≥ 20% in pMMS composite RBS and SFS
Proportion of patients with clinical remission | Weeks 12, 24, 36, 52
  Clinical remission is defined as a pMMS ≤ 2 points, with no individual subscores > 1 point.
Proportion of patients with steroid-free symptomatic remission (among all patients and among patients in symptomatic remission) | Weeks 24, 36, 52
  Steroid-free symptomatic remission is defined as patients in symptomatic remission who did not take any corticosteroid treatment for 8 weeks prior to the visit/timepoint
Proportion of patients with steroid-free clinical remission (among all patients and among patients in clinical remission) | Weeks 24, 36, 52
  Steroid-free clinical remission is defined as patients in clinical remission (using a pMMS) who did not take any corticosteroid treatment for 8 weeks prior to the visit/timepoint
Change from baseline in fatigue | Weeks 12, 24, 36, 52
  Change from baseline in the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue score
  Normalization of fatigue is defined as a FACIT Fatigue score ≥ 40.1
Change from baseline of bowel urgency | Weeks 12, 24, 36, 52
  Change from baseline in bowel urgency on a 0 (no urgency) - 10 (worst possible urgency) numeric rating scale
Proportion of patients with a clinically meaningful improvement in bowel urgency | Weeks 12, 24, 36, 52
  Clinically meaningful improvement in bowel urgency is defined as ≥ 3-point decrease from baseline among patients with baseline bowel urgency score ≥ 3
Proportion of patients in bowel urgency remission | Weeks 12, 24, 36, 52
  Bowel urgency remission is defined as a bowel urgency score ≤ 1 among patients with a baseline bowel urgency score ≥ 3 and the overall population
Proportion of patients with complete bowel urgency remission | Weeks 12, 24, 36, 52
  Complete bowel urgency remission is defined as a bowel urgency Numeric Rating Scale score = 0
Change from baseline in abdominal pain | Weeks 12, 24, 36, 52
  Change from baseline in abdominal pain on a 0 (no pain) - 10 (pain as bad as can imagine) numeric rating scale
Proportion of patients with abdominal pain remission | Weeks 12, 24, 36, 52
  Abdominal pain remission is defined as an abdominal pain Numeric Rating Scale score = 0

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Reddy GI Associates, Mesa, Arizona
  - Scripps Clinic Torrey Pines, La Jolla, California
  - United Medical Doctors, Los Alamitos, California
  - Amicis Research Center, Valencia, California
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - Gastro Florida, Lutz, Florida
  - Orlando Health/Digestive Health Institute, Orlando, Florida
  - Best Choice Medical Research Service, Pembroke Pines, Florida
  - University of South Florida, Tampa, Florida
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Woodholme Gastroenterology Associates PA, Glen Burnie, Maryland
  - NYU Langone Health, New York, New York
  - Lenox Hill Hospital, Northwell Health, New York, New York
  - University of North Carolina at Chapel Hill, Division of Gastroenterology and Hepatology, Chapel Hill, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, LLC, Westlake, Ohio
  - Houston Endoscopy & Research Center, Houston, Texas
  - BI Research Center, Houston, Texas
  - Brooke Army Medical center, San Antonio, Texas
  - GI Alliance Research, Southlake, Texas
  - Washington Gastroenterology, Tacoma, Washington
  - WVU Medicine J.W Ruby Memorial Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5041047